CLINICAL TRIAL: NCT07296627
Title: A Prospective Study for Chinese Newly Diagnosed Multiple Myeloma Patients Treated With Immuno-therapy in Real-world Setting
Brief Title: Real-world Immuno-therapy in Chinese Newly Diagnosed Multiple Myeloma Patients
Acronym: PRIMARY
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Dr, Peking University People's Hospital
Other Study IDs: 2024PHB463-001
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Newly Diagnosed Multiple Myeloma (NDMM)
Keywords: Immuno-therapy; anti-CD38 monoclonal antibodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed multiple myeloma

SUMMARY:
To conduct a multicenter, prospective observational cohort study to investigate first-line immunotherapy patterns and clinical outcomes in NDMM patients in China. Leveraging the extensive patient resources of China's large center for blood disorders, the investigator will recruit approximately 500 NDMM patients to establish an NDMM patient cohort. The investigator will collect data on disease characteristics, treatment patterns, and clinical outcomes through one year of clinical follow-up. Further long-term follow-up is needed to obtain survival status and causes of death, so as to provide essential evidence for optimizing and improving patients' prognosis in clinical individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma (NDMM)
* Plan to receive first-line immunotherapy at the respective research center
* First-line immunotherapy includes proteasome inhibitors (PI), immunomodulatory drugs (IMiDs), or anti-CD38 monoclonal antibodies, used alone or in combination with each other or with other treatments
* Age ≥ 18 years
* Ability to understand the purpose of the study and follow-up process
* Willingness to provide signed and dated written informed consent

Exclusion Criteria:

- Patients who did not receive any follow-up after initial diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: it is expected that approximately 500 newly diagnosed multiple myeloma patients will be able to participate in the study during the study period of the selected centers.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
treatment patterns | From July 2025 to July 2026
  To describe the treatment patterns of Chinese NDMM patients receiving first-line immunotherapy in real-world settings.
real-world overall response rate (rwORR) | From July 2025 to July 2026
  To determine the clinical outcomes of Chinese NDMM patients receiving first-line immunotherapy in real-world settings.The real-world overall response rate (rwORR) of the entire population, as well as the rwORR of each treatment regimen.

SECONDARY OUTCOMES:
MRD | July 2025-July 2027
  To assess the depth of response in Chinese patients with NDMM receiving first-line immunotherapy in real-world settings, with the corresponding endpoint being minimal residual disease.
Revised International Staging System (R-ISS) Stage | July 2025-July 2026
  Disease stage classified according to the Revised International Staging System (R-ISS I, II, or III) at baseline.
Serum Lactate Dehydrogenase Level | July 2025-July 2026
  Serum LDH concentration measured at baseline, reported in units per liter (U/L).
Age at Baseline | July 2025-July 2026
  Patient age in years at the time of enrollment (baseline)
Sex | July 2025-July 2026
  Biological sex recorded at baseline (male or female)
M-Protein Isotype | July 2025-July 2026
  Type of monoclonal immunoglobulin (e.g., IgG, IgA, IgD, IgM, light chain only) determined at diagnosis.
Gain of Chromosome 1q21 by FISH | July 2025-July 2026
  Presence of gain or amplification of chromosome region 1q21 detected by FISH at baseline
Ultra-High-Risk Cytogenetic Abnormalities (UHRCA) | July 2025-July 2026
  Presence of ultra-high-risk genetic features defined as: TP53 biallelic inactivation, ≥2 high-risk cytogenetic lesions (e.g., del(17p), t(4;14), amp(1q)), circulating plasma cells ≥2%, or primary refractory disease

CONTACTS AND LOCATIONS:
Overall Officials: Prof. LU, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No